CLINICAL TRIAL: NCT03249181
Title: Dolutegravir in Pregnant HIV Mothers and Their Neonates
Acronym: DolPHIN-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: UNITAID (Other); University of Cape Town (Other); Liverpool School of Tropical Medicine (Other); Infectious Diseases Institute, Uganda (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DolPHIN-2
Record Dates: First submitted 2017-07-28; First posted 2017-08-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2023-11

CONDITIONS: HIV-1-infection; Pregnancy Related
Keywords: MTCT; Antiretroviral; Pregnancy; Africa
MeSH Terms: interventions — dolutegravir; Standard of Care; efavirenz

STUDY DESIGN:
Intervention Model Description: An open-label, multi-centre randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dolutegravir (Experimental): Dolutegravir group (DTG+2 NRTIs) - to make best comparison with standard of care, these NRTIs should be those recommended by national policy.
  Participants randomized to the study drug will be commenced on an antiretroviral regimen comprising DTG 50mg once daily in combination with 2 NRTIs
  Interventions: Drug: Dolutegravir
- Standard of Care (EFV + 2 NRTI backbone) (Active Comparator): Participants randomized to receive standard of care will receive the currently used antiretroviral regimens in keeping with national policy (EFV + 2NRTIs at both study sites).
  Interventions: Drug: Standard of Care (EFV + 2 NRTI backbone)

INTERVENTIONS:
Drug: Dolutegravir — Patients randomized to the study drug will be commenced on an antiretroviral regimen comprising DTG 50mg once daily in combination with 2 NRTIs
  Arms: Dolutegravir
Drug: Standard of Care (EFV + 2 NRTI backbone) — Patients randomized to receive standard of care will receive the currently used antiretroviral regimens in keeping with national policy.
  Arms: Standard of Care (EFV + 2 NRTI backbone)

SUMMARY:
To evaluate dolutegravir (DTG) efficacy in women who present with untreated HIV in late pregnancy.

An open-label, multi-centre randomised controlled trial of DTG vs efavirenz-based regimens for women commencing cART in late pregnancy. HIV positive pregnant women presenting with untreated HIV infection in late (≥28 weeks gestation) pregnancy will be randomised 1:1 to receive DTG (50mg once daily) + 2 nucleoside reverse transcriptase inhibitors (NRTIs) or EFV + 2 NRTIs (SoC)

DETAILED DESCRIPTION:
This is an open-label, randomised controlled trial of DTG versus EFV -based regimens for 250 women commencing cART in late pregnancy, randomised 1:1 to DTG vs EFV-based cART. The purpose of this study is to inform treatment guidelines and for the first time specifically address the treatment needs of this group of women- hence the trial is powered for superiority over EFV. The primary endpoints is maternal VL at delivery, with secondary endpoints including safety and tolerability of DTG in both mother and infant, VL decline in breast milk, development of drug resistance, pharmacokinetics of DTG in mother-infant pairs, pharmacogenomics factors relating to efficacy or toxicity of DTG, and MTCT of HIV up to 72 weeks postpartum. Two sites have been selected - Infectious Diseases Institute, Makerere University, Kampala, Uganda and the University of Cape Town, South Africa - both have a strong track record of successfully delivering collaborative multidisciplinary research in PMTCT. Furthermore, health economics analysis to examine costs and cost-effectiveness of DTG in late-presenting pregnant women will be conducted

The desired outcome of this project is to establish high quality evidence and operational guidance for use of DTG in late pregnancy. Late-presenting HIV-infected pregnant women are an important, but neglected group of vulnerable individuals in whom a randomised controlled intervention of HIV treatment has never previously been undertaken. This work will be done in relationship with WHO and the Clinton Health Access Initiative to ensure successful delivery of the project objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Women aged 18 years or older
4. Pregnant ( ≥28 weeks gestation by best available gestation estimation)
5. Untreated HIV infection in late pregnancy

Exclusion Criteria:

1. Received any antiretroviral drugs in previous 12 months
2. Ever received integrase inhibitors
3. Previous documented failure of an NNRTI-containing ART regimen, previous EFV-associated toxicity or other history of ARV use that would preclude randomisation based on investigator judgement
4. Serum haemoglobin <8.0 g/dl
5. eGFR<50 ml/min*
6. Elevations in serum levels of alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN) or ALT >3xULN and bilirubin >2xULN (with >35% direct bilirubin).
7. History or clinical suspicion of unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hyperbilirubinaemia, oesophageal or gastric varices or persistent jaundice).
8. Severe pre-eclampsia (e.g. HELLP), or other pregnancy related events such as renal or liver abnormalities (e.g. grade 2 or above proteinuria,, total bilirubin, ALT or AST)* at the time of enrolment
9. Paternal objection for infant participation in DTG arm (where disclosure has taken - applies to Uganda site only
10. Medical, psychiatric or obstetric condition that might affect participation in the study based on investigator judgement
11. Receiving any of the following medications (current or within past 2 weeks): anti-epileptic drugs, TB therapy, or other drugs known to significantly interact with either DTG or EFV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
HIV Viral Load at Delivery | by delivery
  <50 copies/ mL

SECONDARY OUTCOMES:
Plasma viral load | By delivery
  <1000 copies/ mL
Maternal viral load to 48 weeks | 48 weeks postpartum
  Proportion <50 and <1000 copies/ mL
Maternal viral load to 72 weeks | 72 weeks postpartum
  Proportion <50 and <1000 copies/ mL
Occurrence of MTCT | 48 weeks postpartum
  Proportion of infants with HIV infection
Occurrence of MTCT | 72 weeks postpartum
  Proportion of infants with HIV infection

OTHER OUTCOMES:
Drug toxicities as defined by DAIDS criteria | Each study visit up to 72 weeks postpartum
  Safety questionnaire
Drug toxicities as defined by DAIDS criteria | Each study visit up to 72 weeks postpartum
  CBC
Drug toxicities as defined by DAIDS criteria | Each study visit up to 72 weeks postpartum
  Serum creatinine (mg/dL)
Drug toxicities as defined by DAIDS criteria | Each study visit up to 72 weeks postpartum
  ALT (U/mL)
Drug toxicities as defined by DAIDS criteria | Each study visit up to 72 weeks postpartum
  Blood urea nitrogen (mg/dL)
Drug toxicities as defined by DAIDS criteria | Each study visit up to 72 weeks postpartum
  Creatine phosphokinase (U/mL)
Safety endpoint: Maternal mental health (Edinburgh Postnatal Depression Scale) | Enrolment, 4 weeks after ART initiation, every postnatal visit up to 72 weeks postpartum
  Edinburgh Postnatal Depression Scale
Safety endpoint: Maternal mental health (Hospital Anxiety and Depression Scale) | Enrolment, 4 weeks after ART initiation, every postnatal visit up to 72 weeks postpartum
  Hospital Anxiety and Depression Scale
Safety of DTG in infant: Birth outcomes (Surface examination for anomalies) | At birth
  Surface examination for anomalies
Safety of DTG in infant: Birth outcomes (Ballard Score for Maturity) | At birth
  Ballard Score for Maturity
Safety of DTG in infant: Birth outcomes (Weight) | At birth
  Weight
Safety of DTG in infant: Birth outcomes (Length) | At birth
  Length
Safety of DTG in infant: Growth and development (Infant gross motor screening tool) | 24, 48 and 72 weeks postpartum
  Infant gross motor screening tool
Safety and tolerability of DTG exposure to infant: Maternal report (Safety questionnaire) | Delivery and all postnatal follow-up to 72 weeks
  Safety questionnaire
Safety of DTG exposure to infant (Blood glucose) | Delivery and 6 weeks postpartum
  Blood glucose
Safety of DTG exposure to infant | 6 weeks postpartum
  ALT (U/mL)
Safety of DTG exposure to infant | 6 weeks postpartum
  Blood urea nitrogen (mg/dL)
Safety of DTG exposure to infant | 6 weeks postpartum
  Serum creatinine (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Saye H Khoo, Study Chair — University of Liverpool
Locations (2):
- University of Cape Town, Cape Town, Western Cape, South Africa
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiiza D, Rostami-Hochaghan D, Alhassan Y, Seden K, Reynolds H, Kaboggoza JP, Taegtmeyer M, Chen T, Challenger E, Malaba T, Wang D, Else L, Hern F, Sharp J, Neary M, Dilly Penchala S, Waitt C, Orrell C, Colbers A, Myer L, Owen A, Rannard S, Khoo S, Lamorde M. Clinical, pharmacological, and qualitative characterization of drug-drug interactions in pregnant women initiating HIV therapy in Sub-Saharan Africa. J Antimicrob Chemother. 2024 Sep 3;79(9):2334-2342. doi: 10.1093/jac/dkae232. PMID 38997229
- [Derived] Malaba TR, Nakatudde I, Kintu K, Colbers A, Chen T, Reynolds H, Read L, Read J, Stemmet LA, Mrubata M, Byrne K, Seden K, Twimukye A, Theunissen H, Hodel EM, Chiong J, Hu NC, Burger D, Wang D, Byamugisha J, Alhassan Y, Bokako S, Waitt C, Taegtmeyer M, Orrell C, Lamorde M, Myer L, Khoo S; DolPHIN-2 Study Group. 72 weeks post-partum follow-up of dolutegravir versus efavirenz initiated in late pregnancy (DolPHIN-2): an open-label, randomised controlled study. Lancet HIV. 2022 Aug;9(8):e534-e543. doi: 10.1016/S2352-3018(22)00173-4. PMID 35905752
- [Derived] Ochanda PN, Lamorde M, Kintu K, Wang D, Chen T, Malaba T, Myer L, Waitt C, Reynolds H, Khoo S. A randomized comparison of health-related quality of life outcomes of dolutegravir versus efavirenz-based antiretroviral treatment initiated in the third trimester of pregnancy. AIDS Res Ther. 2022 Jun 7;19(1):24. doi: 10.1186/s12981-022-00446-3. PMID 35672853
- [Derived] Kintu K, Malaba TR, Nakibuka J, Papamichael C, Colbers A, Byrne K, Seden K, Hodel EM, Chen T, Twimukye A, Byamugisha J, Reynolds H, Watson V, Burger D, Wang D, Waitt C, Taegtmeyer M, Orrell C, Lamorde M, Myer L, Khoo S; DolPHIN-2 Study Group. Dolutegravir versus efavirenz in women starting HIV therapy in late pregnancy (DolPHIN-2): an open-label, randomised controlled trial. Lancet HIV. 2020 May;7(5):e332-e339. doi: 10.1016/S2352-3018(20)30050-3. PMID 32386721